CLINICAL TRIAL: NCT00651586
Title: Safety and Efficacy Study of Gatifloxacin Compared With Ciprofloxacin in Patients With Acute Bacterial Corneal Ulcers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Therapeutic Area Head, Allergan, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 198782-002
Record Dates: First submitted 2008-04-01; First posted 2008-04-03 (Estimated); Last update posted 2008-07-29 (Estimated); Status verified 2008-07

CONDITIONS: Acute Bacterial Corneal Ulcers; Bacterial Keratitis
MeSH Terms: interventions — Gatifloxacin; Ophthalmic Solutions; Ciprofloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental): Gatifloxacin 0.3% ophthalmic solution
  Interventions: Drug: Gatifloxacin 0.3% ophthalmic solution
- 2 (Active Comparator): Ciprofloxacin 0.3% ophthalmic solution
  Interventions: Drug: Ciprofloxacin 0.3% ophthalmic solution

INTERVENTIONS:
Drug: Gatifloxacin 0.3% ophthalmic solution — Gatifloxacin 0.3% ophthalmic solution. On Day 0, one drop instilled in affected eye every 5 minutes for the first 30 minutes, every 30 minutes while awake, and every 2 hours after retiring; on Day 1, one drop instilled in affected eye every hour while awake and 4 hours after retiring; on Days 2 to 6, one drop instilled in affected eye every 2 hours while awake; on Days 7 to 21, one drop instilled in affected eye 4 times daily while awake. Treatment continued through Day 21 (or Day 28 if ulcer had not healed but was improving); dosing terminated when re-epithelialization was complete or on Day 28, whichever occurred sooner
  Arms: 1
Drug: Ciprofloxacin 0.3% ophthalmic solution — Ciprofloxacin 0.3% ophthalmic solution. On Day 0, one drop instilled in affected eye every 5 minutes for the first 30 minutes, every 30 minutes while awake, and every 2 hours after retiring; on Day 1, one drop instilled in affected eye every hour while awake and 4 hours after retiring; on Days 2 to 6, one drop instilled in affected eye every 2 hours while awake; on Days 7 to 21, one drop instilled in affected eye 4 times daily while awake. Treatment continued through Day 21 (or Day 28 if ulcer had not healed but was improving); dosing terminated when re-epithelialization was complete or on Day 28, whichever occurred sooner
  Other Names: Ciloxan®
  Arms: 2

SUMMARY:
This study evaluates the safety and efficacy of gatifloxacin 0.3% ophthalmic solution compared with ciprofloxacin 0.3% ophthalmic solution in patients with acute bacterial corneal ulcers

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis in one eye only of an acute bacterial corneal ulcer (>1mm)

Exclusion Criteria:

* Corneal ulcer that in the opinion of the investigator had to be treated with fortified antibiotics, or multiple antibiotics, or anti-infectives other than study medication

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2003-10; Primary Completion 2005-04 (Actual); Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
Complete re-epithelialization of the corneal ulcer | Day 21

SECONDARY OUTCOMES:
Investigator's evaluation of clinical efficacy | Day 21
Patient reported outcomes | Day 21
Microbiological Cure | Day 21

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (2):
- Galveston, Texas, United States
- Madurai, Tamil Nadu, India

REFERENCES:
- [Background] Prajna V, Vajpayee R, Trocme S, Davitt WF, III, Jensen H, Liu R, Safyan E. Safety and Efficacy of Gatifloxacin 0.3% as Compared With Ciprofloxacin 0.3% for the Treatment of Acute Bacterial Corneal Ulcers. Investigative Ophthalmology & Visual Science. 5-1-2006; 47(5):1916
- See also: Link to Clinical Trial Results — http://www.allerganclinicaltrials.com